CLINICAL TRIAL: NCT07176039
Title: Comparison Between High-Intensity Laser Therapy and Extracorporeal Shockwave Therapy in the Treatment of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, reda abd elrazik, Associate Professor, Department of Physical Therapy for musculoskeletal disorders and its surgery, Faculty of Physical Therapy, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT.BU.EC.23
Record Dates: First submitted 2025-09-01; First posted 2025-09-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Pain Syndrome - Neck
Keywords: Myofascial Pain Syndrome; High-Intensity Laser Therapy; Extracorporeal Shockwave Therapy; Cervical Pain; Physical Therapy; Pain Management
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain; Agnosia | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Laser Therapy (HILT) (Experimental): Participants will receive High-Intensity Laser Therapy (HILT) applied to active myofascial trigger points in the neck and shoulder region, using an 808 nm GaAlAs laser, 8-10 W, 2000 Hz, 60 seconds per point, 5-6 points per session, twice weekly for 4 weeks (8 sessions total).
  Interventions: Radiation: High-Intensity Laser Therapy (HILT)
- Extracorporeal Shockwave Therapy (ESWT) (Active Comparator): Participants will receive Extracorporeal Shockwave Therapy (ESWT) using a radial shockwave device with energy flux density of 0.1-0.2 mJ/mm², 2000 shocks per session, administered twice weekly for 4 weeks (8 sessions).
  Interventions: Other: Extracorporeal Shockwave Therapy (ESWT)

INTERVENTIONS:
Radiation: High-Intensity Laser Therapy (HILT) — will be administered to active myofascial trigger points in the neck and shoulder region. The laser device used is an 808 nm gallium-aluminum-arsenide (GaAlAs) diode laser in continuous mode. Parameters: power output of 8-10 W, frequency of 2000 Hz, and application time of 60 seconds per trigger point, targeting 5-6 trigger points per session. Treatment will be delivered twice weekly for 4 consecutive weeks, totaling 8 sessions.
  Arms: High-Intensity Laser Therapy (HILT)
Other: Extracorporeal Shockwave Therapy (ESWT) — ESWT will be applied to active myofascial trigger points using a radial shockwave device. Parameters: Energy flux density 0.1-0.2 mJ/mm², 2000 shocks per session, frequency of 2 sessions per week for 4 weeks (8 sessions).
  Arms: Extracorporeal Shockwave Therapy (ESWT)

SUMMARY:
this randomized controlled trial aims to compare the effectiveness of High-Intensity Laser Therapy (HILT) and Extracorporeal Shockwave Therapy (ESWT) in managing patients with Myofascial Pain Syndrome (MPS). Thirty-two participants will be randomly assigned to receive either HILT or ESWT over a period of 4 weeks. Outcome measures include pain intensity (Visual Analog Scale), tenderness, functional disability, and cervical range of motion.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the efficacy of High-Intensity Laser Therapy (HILT) and Extracorporeal Shockwave Therapy (ESWT) in the management of patients with Myofascial Pain Syndrome (MPS) of the neck and shoulder region. Thirty-two participants will be randomly allocated into two groups: one receiving HILT and the other receiving ESWT, with both groups undergoing 8 treatment sessions over 4 weeks. The primary outcome is pain intensity assessed by the Visual Analog Scale (VAS). Secondary outcomes include tenderness (PPT), functional disability (Neck Disability Index), and cervical range of motion (measured by CROM). The study will be conducted at the Faculty of Physical Therapy, Benha University.

ELIGIBILITY:
Inclusion Criteria:

Male and female participants aged 18-60 years. Diagnosis of Myofascial Pain Syndrome (MPS) in the neck/shoulder region. Presence of active myofascial trigger points in the upper trapezius. Willingness to provide informed consent.

Exclusion Criteria:

History of cervical spine surgery, trauma, or radiculopathy. Contraindications to laser or shockwave therapy. Presence of systemic diseases (e.g., rheumatoid arthritis, malignancy). Receiving other physical therapy interventions during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Pain Intensity | Baseline and 4 weeks after intervention (post-treatment)
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10-cm line where 0 = "no pain" and 10 = "worst pain imaginable". A lower score indicates improvement. The primary outcome is the mean change from baseline to post-treatment.

SECONDARY OUTCOMES:
Pressure Pain Threshold (PPT) as measured by pressure algometer | Baseline and 4 weeks post-treatment
  The pressure pain threshold (PPT) will be assessed using a digital pressure algometer (in kg/cm² or kPa) applied perpendicularly to active myofascial trigger points in the upper trapezius. The point at which the sensation changes from pressure to pain is recorded. Higher values indicate increased pain tolerance. Measurements will be taken at baseline and post-treatment.
Neck Disability Index (NDI) | Baseline and 4 weeks post-treatment
  Functional disability will be assessed using the Neck Disability Index (NDI), a 10-item self-reported questionnaire scored from 0 to 50, where higher scores indicate greater disability. The primary metric is the mean change from baseline to post-treatment.
Cervical Range of Motion (ROM) | Baseline, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: reda K. Abdelrazik, associate professor, Principal Investigator — Benha University
Locations (1):
- Faculty of Physical Therapy, Benha University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No